CLINICAL TRIAL: NCT04703010
Title: Neonatal Precursors of Neurodevelopment
Acronym: NEOPRENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A02117-32
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Magnetic Resonance Imaging; Psychometrics

STUDY DESIGN:
Intervention Model Description: Longitudinal study with measures at birth and at age 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants undergo the same measurements (longitudinal design)
  Interventions: Device: Electroencephalography-Near infrared spectroscopy; Device: Magnetic resonance imaging; Behavioral: Psychometric testing

INTERVENTIONS:
Device: Electroencephalography-Near infrared spectroscopy — Brain activity will be measured using 128-channel EEG and 2 channel NIRS during tactile stimulation (15 minutes sequence of vibrations) while the newborn is asleep.
Device: Magnetic resonance imaging — Structural (T1-T2), siffusion tensor imaging and blood-oxygen level dependant signal will be acquired in a subset of 40 subjects (20 minutes while asleep)
Behavioral: Psychometric testing — Cognitive evaluation at age 2 (Parental questionnaires on sensory profiles, executive functions and neurodevelopmental disorders screening, child tests : movement assessment battery, Laby, Head-toes-shoulders-knees)

SUMMARY:
The NEOPRENE project proposes to examine processes that are among the earliest precursors of cognitive functions and assess 1) the relationship between neonatal cognitive precursors and cortical structure, structural connectivity and functional connectivity at birth and 2) the relationship between neonatal cognitive precursors and neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborn (born < 34 weeks + 6days)

Exclusion Criteria:

* Brain injury
* Respiratory assistance on measurement day
* Infection on measurement day
* Sedation on measurement day
* Parents < 18 years old or unable to give informed consent

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography evoked response amplitude | 35 weeks of gestational age
  Electrical field potential changes in the parietal and frontal cortices
Near infrared spectroscopy evoked response amplitude | 35 weeks of gestational age
  Oxygenated hemoglobin concentration changes in the somatosensory cortex
Grey matter volume in the somatosensory cortex | 35 weeks GA
  Thickness measured on T2 images in magnetic resonance imaging
Frontal-parietal structural connectivity | 35 weeks GA
  Tractography using Diffusion tensor Imaging in magnetic resonance imaging
Frontal-parietal functional connectivity | 35 weeks GA
  Synchronization at rest using blood-oxygen level dependent signal in magnetic resonance imaging
Quality of cognitive development | 2 years old
  Qualitative composite assessment using clinical interview, routine pediatric screening and questionnaires (full sensory profile, preschooler Behavior Rating Inventory of Executive Function)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: funding information — https://anr.fr/Projet-ANR-19-CE37-0015